CLINICAL TRIAL: NCT03425682
Title: A Prospective, Post-Market, Multi-Center Study Evaluating ViBone® in Cervical and Lumbar Spine Fusion
Brief Title: ViBone in Cervical and Lumbar Spine Fusion
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0001
Record Dates: First submitted 2018-01-29; First posted 2018-02-07 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Spondylosis; Cervical Spondylosis; Spondylolisthesis; Herniated Nucleus Pulposus; Degenerative Disc Disease
Keywords: Anterior Cervical Discectomy and Fusion (ACDF); Transforaminal Lumbar Interbody Fusion (TLIF); Posterior Lumbar Interbody Fusion (PLIF)
MeSH Terms: conditions — Spondylosis; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical Fusion - ACDF: Patients undergoing anterior cervical discectomy and fusion (ACDF) using ViBone will be enrolled.
  Interventions: Other: ViBone
- Lumbar Interbody Fusion: Patients undergoing lumbar interbody fusion (TLIF, PLIF, ALIF, or LLIF) using ViBone will also be enrolled.
  Interventions: Other: ViBone

INTERVENTIONS:
Other: ViBone — Viable Bone Allograft

SUMMARY:
Assess clinical and radiographic outcomes in patients who undergo 1-3 level anterior cervical discectomy fusion (ACDF) or lumbar interbody fusion (TLIF, PLIF, ALIF, or LLIF) using ViBone.

DETAILED DESCRIPTION:
This study is a prospective, multi-center study to evaluate the clinical and radiographic outcomes of ViBone in patients undergoing ACDF or lumbar interbody fusion. Data will be gathered for subjects undergoing ACDF surgery and subjects undergoing lumbar fusion surgery using ViBone. Total enrollment is expected to be approximately 100 subjects. The purpose of this study is to assess clinical and radiographic outcomes in patients who undergo 1-3 level ACDF or lumbar interbody fusion surgery using ViBone. Subjects will be followed for 12 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-80 years of age
* For cervical cases - ACDF surgery at 1, 2, or 3 contiguous levels between C2-C7
* For lumbar cases - lumbar interbody fusion surgery at 1, 2, or 3 contiguous levels between L1-S1
* Patient signed Consent Form with HIPAA Authorization
* Appropriate candidate for surgery
* Patient will adhere to the scheduled follow-up visits and requirements of the protocol including routine patient exams - pre-operative, operative, and at least two post- operative visits (6 and 12 months post-surgery). Pre-operative and post-operative visits include X-ray (required) and CT scan (if available).

Exclusion Criteria:

* Long term use of medications that are known to inhibit fusion or bone metabolism or immune suppressants 6 months prior to surgery (i.e., steroids, chemotherapy, DMARDs, etc.)
* Treatment with radiotherapy
* Acute or chronic systemic or localized spinal infections
* Instability associated with major reconstructive surgery for primary tumors or metastatic malignant tumors of the cervical (for ACDF patients) or lumbar (for TLIF, PLIF, ALIF, or LLIF patients) spine
* Previous pseudoarthrosis at any level of the cervical (for ACDF patients) or lumbar (for
* TLIF, PLIF, ALIF, or LLIF patients) spine
* Nursing mothers or women who are pregnant or plan to become pregnant during the course of the study
* Current or recent history of malignancy or infectious disease. Patients with current or recent history of basal cell carcinoma are eligible.
* Inability to provide informed consent
* Rapid joint disease, bone absorption, osteomalacia, and/or diagnosed osteoporosis (bone density score of ≤-2.5).
* Other medical or surgical conditions which would preclude the potential benefit of surgery, such as congenital abnormalities, immunosuppressive disease, elevation of sedimentation rate unexplained by other diseases, elevation of white blood count (WBC), or marked left shift in the WBC differential count.
* Active local or systemic infection or is undergoing adjunctive treatment for local or systemic infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients, 18-80 years of age undergoing 1-3 level anterior cervical discectomy fusion (ACDF), or lumbar interbody fusion (TLIF, PLIF, ALIF, or LLIF) using ViBone.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Spine Institute of San Diego, San Diego, California
  - Connecticut Neck & Back Specialists, LLC, Danbury, Connecticut
  - Anne Arundel Medical Group, Annapolis, Maryland
  - Orthopedic Specialists of Austin, Austin, Texas

REFERENCES:
- [Derived] Kim PD, Raiszadeh R, Bomback DA, Kramer DL, Moghimi M. 12-Month clinical and radiographic outcomes of ViBone viable bone matrix in patients undergoing cervical and lumbar spinal fusion surgery. J Orthop Surg Res. 2023 Mar 25;18(1):239. doi: 10.1186/s13018-023-03686-9. PMID 36964582

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion
Started | 54 | 64
Completed | 48 | 47
Not Completed | 6 | 17
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Subject did not meet I/E | 4 | 10

BASELINE CHARACTERISTICS:
Population: 95 patients (48 cervical; 47 lumbar) were included in the data analyses because they met the inclusion criteria and had at least one follow-up (6- and/or 12-month).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.1) | 57.8 (9.5) | 56.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 25 | 23 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 25 | 35 | 60
  Race/Ethnicity: Hispanic or Latino | 15 | 10 | 25
  Race/Ethnicity: Black or African American | 4 | 2 | 6
  Race/Ethnicity: Other | 4 | 0 | 4
BMI, Continuous [Mean (Standard Deviation); unit: kg/m²] | 27.9 (5.7) | 29.8 (5.2) | 28.8 (5.5)
BMI, Categorical [Count of Participants; unit: Participants]
  Normal (18.5 - <25.0) | 15 | 6 | 21
  Overweight (25.0 - <30.0) | 17 | 25 | 42
  Obese (30.0 - <40.0) | 16 | 14 | 30
  Morbidly Obese (>/=40.0) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Fusion Rates Per Level Using the Bridwell Interbody Grading Scale
Description: Successful fusion rates for ViBone as defined by Grade I or II level of fusion on the Bridwell Interbody Grading Scale (below). The percentages below show at 12 months the amount of fusion per level for cervical and lumbar fusion procedures utilizing ViBone.
  Grade I: Fused with remodeling and trabeculae present. Grade II: Graft intact, not fully remodeled and incorporated, but no lucency present.
  Grade III: Graft intact, potential lucency present at top and bottom of graft. Grade IV: Fusion absent with collapse/resorption of graft.
Time Frame: 12 months
Population: Subjects with 12 month fusion by level data available
Measure: Count of Units; unit: Fusions
Units Other Than Participants: Fusions
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion
Number analyzed (Participants) | 33 | 25
Number analyzed (Fusions) | 65 | 50
Fusions | 64 | 50

2. Secondary Outcome: Percent Change From Baseline in Oswestry Disability Index (ODI) at 12 Months
Description: Oswestry Disability Index (ODI) improvement relative to baseline for lumbar spine fusion (0-100) 0 is no disability and 100 is bed-bound.
Time Frame: Baseline and 12 months
Population: ODI is not applicable to the cervical fusion arm. 25 subjects had baseline and 12 months data for ODI in the lumbar fusion arm.
Measure: Mean (Standard Deviation); unit: Percent change in ODI from baseline
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion
Number analyzed (Participants) | 0 | 25
Percent change in ODI from baseline |  | -50.6 (55.9)

3. Secondary Outcome: Percent Change From Baseline in Neck Disability Index (NDI) at 12 Months
Description: Neck Disability Index (NDI) improvement relative to baseline for cervical spine fusion Scale of 0 - 100, where 0 is no problems at all and 100 is severely affected.
Time Frame: Baseline and 12 months
Population: NDI is not applicable to the lumbar fusion arm. 33 subjects had NDI data at baseline and 12 months in the cervical fusion arm.
Measure: Mean (Standard Deviation); unit: Percent change in NDI from baseline
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion
Number analyzed (Participants) | 33 | 0
Percent change in NDI from baseline | -41.9 (35.2) |

4. Secondary Outcome: Percent Change From Baseline in Visual Analog Scale (VAS) at 12 Months
Description: Visual Analog Scale (VAS) for pain improvement relative to baseline (Pain scale from 0-10, with 0 being No Pain and 10 being Worst Pain)
Time Frame: Baseline and 12 months
Population: VAS-pain scores were available at baseline and 12 months for 33 subjects in the cervical fusion arm and 25 subjects in the lumbar fusion arm.
Measure: Mean (Standard Deviation); unit: Percent Change from baseline
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion
Number analyzed (Participants) | 33 | 25
Percent Change from baseline | -40.1 (41.5) | -57.5 (44.2)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for up to 1 year.
Arm/Group | Cervical Fusion - ACDF | Lumbar Interbody Fusion
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03425682/Prot_SAP_000.pdf